CLINICAL TRIAL: NCT04894669
Title: Convenience Sample Data Collection for INVSENSOR00045
Status: Terminated | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHOC0006
Record Dates: First submitted 2021-03-17; First posted 2021-05-20 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-02

CONDITIONS: Oxygen Saturation
Keywords: Oxygen Saturation; SpO2

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- INVSENSOR00045 (Experimental): All subjects are enrolled into the test group and are fitted with a non-invasive pulse oximetry sensor called INVSENSOR00045 during their stay at the hospital.
  Interventions: Device: INVSENSOR00045

INTERVENTIONS:
Device: INVSENSOR00045 — Noninvasive sensor will be fitted to the subject's hand, foot, or toe to measure oxygen saturation and pulse rate.

SUMMARY:
This clinical investigation is to collect data to provide additional support for form, fit, and function of INVSENSOR00045 in the neonatal clinical environment when used by hospital's personnel and reference co-oximeter.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 1 month of age
* Gestational age greater than 23 weeks
* Weight less than or equal to 5 kg
* Subjects with standard of care arterial blood sampling line already in place

Exclusion Criteria:

* Subjects with underdeveloped skin
* Subjects with abnormalities at the planned application sites that would interfere with system measurements
* Subjects with known allergic reactions to foam/rubber products and adhesive tape
* Subjects with axillary arterial lines
* Deformities of the limbs, absence of the feet, severe edema, and other at the discretion of the Principal Investigator

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2023-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Site 2, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00045
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00045
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic, Latino or Spanish Origin | 2
  Hispanic, Latino, or Spanish Origin | 3
  Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Form, Fit and Function of INVSENSOR00045.
Description: To observe form, fit, and function of the INVSENSOR00045 sensors in the neonatal population with convenience sampling in a clinical environment. Data collected using the sensors will be compared to the reference values (RMS).
Time Frame: Up to 8 hours per subject.
Population: Data was obtained from all participants and there were no signal quality issues. The study was terminated early and the sample size was insufficient to statistically compare data collected to the reference values. Hence, the root mean square error (RMS) could not be computed.
Measure: Number; unit: number of issues with form/fit &function
Groups:
- INVSENSOR00045: All subjects are enrolled into the test group and are fitted with a non-invasive pulse oximetry sensor called INVSENSOR00045 during their stay at the hospital.
  INVSENSOR00045: Noninvasive sensor will be fitted to the subject's hand, foot, or toe to measure oxygen saturation.
Arm/Group | INVSENSOR00045
Number analyzed (Participants) | 7
number of issues with form/fit &function | 0

ADVERSE EVENTS:
Time Frame: Up to 8 hours
Description: Definitions do not differ.
Arm/Group | INVSENSOR00045
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT04894669/Prot_SAP_000.pdf